CLINICAL TRIAL: NCT06616597
Title: Phase II Trial Targeting Gut Bacterial Androgen Production to Reverse Therapeutic Resistance to Abiraterone in Patients With Metastatic Prostate Cancer
Brief Title: Trial Targeting Gut Bacterial Androgen Production to Reverse Therapeutic Resistance to Abiraterone in Patients With Metastatic Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Prostate Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2485; IRB00453879 (Other: JHM IRB)
Record Dates: First submitted 2024-09-23; First posted 2024-09-27 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer (Adenocarcinoma); Metastatic Prostate Cancer
Keywords: Abiraterone; microbiome; Dexamethasone
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — Abiraterone Acetate; Dexamethasone; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Abiraterone + Dexamethasone (Experimental): Abiraterone acetate plus dexamethasone
  Interventions: Drug: Abiraterone acetate; Drug: Dexamethasone
- Arm 2: Abiraterone + Dexamethasone + metronidazole (Experimental): Abiraterone acetate plus dexamethasone plus metronidazole
  Interventions: Drug: Abiraterone acetate; Drug: Dexamethasone; Drug: Metronidazole

INTERVENTIONS:
Drug: Abiraterone acetate — Abiraterone acetate 1000mg/ day
Drug: Dexamethasone — Dexamethasone 0.5mg/day
Drug: Metronidazole — Metronidazole 1500mg/ per day
  Other Names: Flagyl
  Arms: Arm 2: Abiraterone + Dexamethasone + metronidazole

SUMMARY:
To determine if dexamethasone or dexamethasone plus metronidazole restore sensitivity to abiraterone for the treatment of metastatic prostate cancer.

DETAILED DESCRIPTION:
To test whether giving dexamethasone with or without metronidazole in combination with abiraterone could help reverse resistance to abiraterone for patients with metastatic castration-resistant prostate cancer (mCRPC). Abiraterone and prednisone (AA/P) is a second-line therapy for mCRPC given when first-line androgen deprivation therapy fails. However, resistance to AA/P can develop. The investigators do not know exactly how cancer becomes resistant, but there is evidence that suggests it could be due to androgen production by the bacteria in your gut (gut microbiome). This study is focused on the gut microbiome as a source of androgen production that could cause AA/P resistance in mCRPC.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18 years of age and above.
* Prostate adenocarcinoma
* Absolute PSA ≥ 2.0 ng/mL at screening.
* PSA (+/- radiographic) progression after having been on abiraterone and prednisone for at least 12 weeks.
* Must be maintained on a GnRH analogue or have undergone orchiectomy.
* Participants must have a life expectancy ≥ 6 months
* Ability to swallow study medication tablets
* Willing to abstain from alcohol during and for 14 days after treatment with metronidazole
* Willing and able to collect urine and stool samples per protocol

Exclusion Criteria:

* Active infection or other medical condition that would make dexamethasone use contraindicated
* Any chronic medical condition requiring a higher systemic dose of corticosteroid
* Pathological finding consistent with small cell carcinoma of the prostate
* Has imminent or established spinal cord compression based on clinical findings and/or MRI.
* Chronic liver disease with Child-Pugh class C cirrhosis (see calculator in protocol)
* Bilirubin >3x ULN or AST and ALT >5x ULN
* Congenital prolonged QTc syndrome or QTc > 500 msec (non-paced rhythm)
* History of pituitary or adrenal dysfunction
* Uncontrolled diabetes (Hemoglobin A1c > 10%) or increasing doses of insulin within the past 4 weeks due to poorly controlled glucoses.
* Administration of an investigational therapeutic or invasive surgical procedure (not including surgical castration) within 30 days of Cycle 1 Day 1 or currently enrolled in an investigational drug study
* Any other serious illness or medical condition that would, in the opinion of the investigator, make this protocol unreasonably hazardous, including, but not limited to:

  * Any uncontrolled major infection.
  * Crohn's disease or ulcerative colitis.
  * Known or suspected toxic megacolon and/or known small bowel ileus.
  * Known allergy to any of the compounds under investigation.
* On antibacterial therapy within 30 days prior to administration of study treatment.
* Any condition or situation which, in the opinion of the investigator, would put the subject at risk, or interfere with the subject's participation in this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2031-03-30 (Estimated); Study Completion 2032-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with PSA30 response | 24 weeks
  Number of participants with castration resistant prostate cancer who have a ≥ 30% decline in PSA from baseline until 24 weeks.

SECONDARY OUTCOMES:
Number of participants with PSA50 response | 12 weeks
  Number of participants with castration resistant prostate cancer who have a ≥ 50% decline in PSA from baseline until 12 weeks.
PSA Progression Free Survival | 12 weeks
  Number of participants with PSA progression according to PCWG3 (25% rise in PSA from nadir and increase of at least 2ng/mL)
Number of participants with progression | 24 weeks
  progression is defined as:
  * Progression of soft tissue lesions according to RECIST 1.1 Criteria.
  * Progression of bone lesions detected with bone scan according to PCWG3 criteria.
  * Radiologically-confirmed spinal cord compression or pathological fracture due to malignant progression, or other clinical event deemed to be cancer-related, or death.
Number of grade 3-5 toxicities | 24 weeks
  Toxicity is evaluated based on current CTCAE standard grading scales.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Handy-Marshall, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No